CLINICAL TRIAL: NCT01303536
Title: Ondansetron Augmentation in Treatment-resistant OCD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Neuroscience, Florence, Italy (Other)
Responsible Party: Stefano Pallanti, University of Florence
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: OND2
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Obsessive Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- obsessive compulsive disorder (Experimental): obsessive compulsive patients resistant to selective serotonin reuptake inhibitor therapy, in addition to their continued stable dose of FDA approved selective serotonin reuptake inhibitors, received oral ondansetron 0.25 mg in two daily administrations (0.5 mg daily) for 2 weeks. Subsequently, the dose was titrated to 0.5 mg in two daily administrations (1 mg/day total) for another 10 weeks. ondansetron was discontinued and the patients were followed for an additional 4 week with biweekly
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Ondansetron — obsessive compulsive patients resistant to selective serotonin reuptake inhibitor therapy, in addition to their continued stable dose of FDA approved selective serotonin reuptake inhibitors, received oral ondansetron 0.25 mg in two daily administrations (0.5 mg daily) for 2 weeks. Subsequently, the dose was titrated to 0.5 mg in two daily administrations (1 mg/day total) for another 10 weeks. ondansetron was discontinued and the patients were followed for an additional 4 week with biweekly

SUMMARY:
The aim of this study is to evaluate whether ondansetron augmentation to SSRI will improve and ondansetron discontinuation will result in worsening of obsessive compulsive symptoms among obsessive compulsive disorder resistant patients.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of OCD established by clinical interview with a licensed psychiatrist;
* a score of ≥ 24 at the Yale Brown Obsessive Compulsive Scale
* a Clinical Global Inventory score ≥ 4, after over 12 weeks of treatment with an adequate trial of an selective serotonin reuptake inhibitor at a moderate to high dose

Exclusion Criteria:

* diagnoses of schizophrenia, schizoaffective disorder, organic mental disorder, bipolar disorder, current substance dependence or abuse, and current major depressive episode preceding the onset of obsessive compulsive disorder
* undergoing concomitant behavior therapy
* or having significant cardiovascular, hepatic, renal or pulmonary diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2009-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Yale Brown Obsessive Compulsive Scale | baseline
Yale Brown Obsessive Compulsive Scale | week 2
Yale Brown Obsessive Compulsive Scale | week 4
Yale Brown Obsessive Compulsive Scale | week 6
Yale Brown Obsessive Compulsive Scale | week 8
Yale Brown Obsessive Compulsive Scale | week 10
Yale Brown Obsessive Compulsive Scale | week 12
Yale Brown Obsessive Compulsive Scale | week 14
Yale Brown Obsessive Compulsive Scale | week 16

SECONDARY OUTCOMES:
The Drug Effect scale | week 0
The Drug Effect scale | week 2
The Drug Effect scale | week 4
The Drug Effect scale | week 6
The Drug Effect scale | week 8
The Drug Effect scale | week 10
The Drug Effect scale | week 12
The Drug Effect scale | week 14
The Drug Effect scale | week 16

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Pallanti, MD, Principal Investigator — University of Florence
Locations (1):
- Institute of Neuroscience, Florence, Florence, Italy